CLINICAL TRIAL: NCT02576561
Title: Phase 2a Double-Blind, Randomized, Parallel Group, Dose-Ranging Study to Assess the Safety and Efficacy of Three Doses of TVGV-1 Vaccine Compared to Its Adjuvant, GPI-0100, in Subjects With Histologically Confirmed HPV Induced Cervical HSIL
Brief Title: Safety and Efficacy Study of TVGV-1 Vaccine to Treat HPV Induced Cervical HSIL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: THEVAX Genetics Vaccine (Industry)
Collaborators: Clinical Research Management, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VAX 02-01
Record Dates: First submitted 2015-10-09; First posted 2015-10-15 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Human Papillomavirus; High-Grade Squamous Intraepithelial Lesions
Keywords: human papillomavirus; Cervical Intraepithelial Neoplasia; Cold Knife Conization; hysterectomy; Loop Electrosurgical Excision Procedure; LEEP; HSIL; High-Grade Squamous Intraepithelial Lesion
MeSH Terms: conditions — Squamous Intraepithelial Lesions; Uterine Cervical Dysplasia | interventions — GPI0100; Antigens; Adjuvants, Pharmaceutic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- TVGV-1 (cohort 1) (Experimental): Antigen + Adjuvant - 0.6 mg lyophilized PEK fusion protein + 0.6 ml* GPI- 0100 (1:1 ratio)
  Interventions: Biological: TVGV-1
- GPI-0100 (cohort 1) (Active Comparator): Adjuvant Alone - 0 mg lyophilized PEK fusion protein. 0.6 mg lyophilized placebo cake + 0.6 ml* GPI- 0100 (1:1 ratio)
  Interventions: Biological: GPI-0100
- Placebo (cohort 1) (Placebo Comparator): Placebo- 0 mg lyophilized PEK fusion protein. 0.6 mg lyophilized placebo cake + 0.6 ml placebo-diluent (1:1 ratio)
  Interventions: Biological: Placebo
- TVGV-1 (cohort 2) (Experimental): Antigen + Adjuvant - 0.9 mg lyophilized PEK fusion protein + 0.9 ml* GPI- 0100 (1:1 ratio)
  Interventions: Biological: TVGV-1
- GPI-0100 (cohort 2) (Active Comparator): Adjuvant Alone - 0 mg lyophilized PEK fusion protein. 0.9 mg lyophilized placebo cake + 0.9 ml* GPI- 0100 (1:1 ratio)
  Interventions: Biological: GPI-0100
- Placebo (cohort 2) (Placebo Comparator): Placebo - 0 mg lyophilized PEK fusion protein. 0.9 mg lyophilized placebo cake + 0.9 ml placebo diluent (1:1 ratio)
  Interventions: Biological: Placebo
- TVGV-1 (cohort 3) (Experimental): Antigen + Adjuvant - 1.2 mg lyophilized PEK fusion protein + 1.2 ml* GPI- 0100 (1:1 ratio)
  Interventions: Biological: TVGV-1
- GPI-0100 (cohort 3) (Active Comparator): Adjuvant Alone - 0 mg lyophilized PEK fusion protein + 1.2 mg lyophilized placebo cake 1.2 ml* GPI- 0100 (1:1 ratio)
  Interventions: Biological: GPI-0100
- Placebo (cohort 3) (Placebo Comparator): Placebo - 0 mg lyophilized PEK fusion protein. 1.2 mg lyophilized placebo cake + 1.2 ml placebo-diluent (1:1 ratio)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: TVGV-1 — Antigen + Adjuvant
  Other Names: lyophilized PEK fusion protein; GPI-0100; Antigen; Adjuvant
  Arms: TVGV-1 (cohort 1); TVGV-1 (cohort 2); TVGV-1 (cohort 3)
Biological: GPI-0100 — Adjuvant Alone
  Other Names: Adjuvant
  Arms: GPI-0100 (cohort 1); GPI-0100 (cohort 2); GPI-0100 (cohort 3)
Biological: Placebo — Placebo
  Other Names: lyophilized placebo cak; placebo diluent; sterile water
  Arms: Placebo (cohort 1); Placebo (cohort 2); Placebo (cohort 3)

SUMMARY:
The purpose of this research study is to test the safety and effectiveness of the investigational study vaccine, called TVGV-1. The study will test the vaccine in women with high grade HPV cervical infection.

DETAILED DESCRIPTION:
The purpose of the Phase 2a Study VAX 02-01 is to assess the safety and activity of TVGV-1 vaccine construct in achieving the absence of histologic HSIL (CIN2/3) (regression to LSIL or less) as assessed by biopsy at last study Visit 11, Day 270.

The objective of the TVGV-1 program is to develop a non-surgical alternative that is reliable, safe, and would avoid potential surgical risks such as preterm birth, perinatal mortality, risk of infertility, incontinence and disfigurement, as well as reduced cost and inconvenience for an otherwise economically productive young subject population.

ELIGIBILITY:
Inclusion Criteria:

1. Female age 18 to 55 years
2. Written informed consent in accordance with institutional guidelines
3. Negative pregnancy test (urine and blood tests)
4. Women of child bearing potential must agree to use contraception through one menstrual cycle post end of study or if early withdrawal, through what would have been visit 11. Methods include intrauterine device or double barrier method, hormonal contraceptive in combination with a double barrier method.
5. Patients who have ONLY HPV 16 OR HPV 16 AND 18 and no other High-Risk HPV by Cobas test will be included.
6. Histologically confirmed, positive HSIL of CIN2+ or higher (only CIN2+/3 subjects will be selected) cervical biopsy, confirmed by external (independent) pathologist panel within the 12 weeks prior to enrollment. If the standard care biopsy is not available for evaluation by the independent pathologist, a fresh biopsy and endocervical curettage will be required. The extent of colposcopic HSIL disease should not involve more than two quadrants of the cervix. Biopsies should be taken from each affected quadrant
7. Adequate visualization of entire cervix, cervical lesion(s) and squamous-columnar junction
8. Normal electrocardiogram (ECG), laboratory values (chemistry, complete blood count) and urinalysis, as judged Grade 0-1 by per National Cancer Institute Common Toxicity Criteria (NCI-CTC)
9. Agrees to Loop Electrosurgical Excision Procedure (LEEP), Cold Knife Conization (CKC) or Hysterectomy being performed at the end of study according to the standard-of-care

Exclusion Criteria:

1. History of cancer (excluding basal cell carcinoma of the skin) including cervical cancer
2. Eastern Cooperative Oncology Group (ECOG) performance status >2 (See Appendix G)
3. Administration of any blood product within 3 months of enrollment
4. Active infection requiring antimicrobial treatment that would interfere with interpretation of adverse events, cutaneous reactions or efficacy. Treatment of minor concurrent infections should be limited to less than 10 days.
5. Administration of any vaccine within 8 weeks of enrollment and within 4 weeks for flu vaccine.
6. Participation in any study with an investigational compound or device within 30 days prior to signing informed consent
7. Any hematologic disorder involving platelets or clotting abnormalities or any condition requiring treatment with transfusions, anticoagulants except platelet inhibitors (NSAIDs as needed for pain are permitted)
8. Active drug or alcohol use or dependence that, in the opinion of the Site Investigator, would interfere with adherence to study protocol
9. Skin conditions that require consistent use of topical corticosteroids or other local or systemic therapy that may interfere with interpretation or description of skin-related adverse events linked to vaccination
10. The standard criteria for prospective clinical trials of medications developed by Drug-Induced Liver Injury Network (established by The National Institute of Diabetes and Digestive and Kidney Diseases) will be used to assess the laboratory test abnormalities. Normal range for these labs will typically be 5 - 40 IU/L for AST; 7 - 56 IU/L for ALT; 0.2 - 1.2 mg/dL for bilirubin. Subjects will be excluded if values are x 2-x 2.5 the upper limit
11. Evidence of hematopoietic, cardiovascular, hepatic, renal, neurologic, psychiatric, dermatologic, immune disorder, or other disease that may interfere with assessment of safety or efficacy of vaccine activity as indicated in study objectives
12. Any known allergic reaction to vaccine components
13. Any other medical condition(s) that, in the judgment of the Site Investigator, might interfere with the study or require treatment that might interfere with the study
14. Family member of the investigation study staff
15. Pregnant or breast-feeding
16. Inability to provide informed consent
17. A subject with a history or expectation of noncompliance with medications or treatment protocol
18. Receipt of (e.g. Gardasil® or Cervarix®) HPV preventative vaccines within 8 years of study enrollment
19. Excessive use of acetaminophen or other potentially hepatotoxic drugs

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-11; Primary Completion 2018-05 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Absence of histologic HSIL (CIN2/3) as assessed by biopsy at last study Visit 11, Day 270. | DAY 270
  The primary analysis for efficacy will be a comparison between subjects treated with and without the PEK fusion protein with respect to the percentage who present regression of HSIL at Day 270. Separate comparisons within each cohort will be performed using Fisher's exact test (or an appropriate analogue). No adjustment for multiple comparisons will be employed in these analyses. Additionally, a corresponding comparison across all study subjects combined will be performed, based on Cochran-Matel-Haenszel test stratified for cohort.
Assessment of cutaneous toxicities (i.e., size, induration and time to resolution of skin reactions to vaccine). | DAY 270
  Summaries of the data pertaining to the primary safety outcome of skin toxicity will be provided. Summaries will be provided for the within-cohort subsets of subjects treated with the active, and with the adjuvant alone; and the combined subsets across all three cohorts of subject treated with the active, with the adjuvant alone, and with the placebo. Serious adverse events will be described in narrative with the participant's demographics, treatment date, event, onset date, relationship to the study treatment and the descriptions of the actions and outcomes during this event. Any deaths occurring in the study will be summarized in narrative with the demographics, treatment duration, cause of death, date of death and additional information surrounding that serious adverse event.

SECONDARY OUTCOMES:
Absence of HPV16 in cervical cytological specimen. Absence of cervical dysplasia 6 months and 8 months after last dose of TVGV-1. | DAY 270
  The primary analysis for efficacy will be a comparison between subjects treated with and without the PEK fusion protein with respect to the percentage who present regression of HSIL at Day 270. Separate comparisons within each cohort will be performed using Fisher's exact test (or an appropriate analogue). No adjustment for multiple comparisons will be employed in these analyses. Additionally, a corresponding comparison across all study subjects combined will be performed, based on Cochran-Matel-Haenszel test stratified for cohort.
Assessment of clinical or laboratory findings and other safety variables. | DAy 270
  Appropriate laboratory data will be transformed prior to analysis as defined in the Statistical Analysis Plan (SAP). Summaries will be presented for each evaluation time point, as well as for changes from baseline. Changes from baseline will also be presented using shift tables for selected laboratory parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Frank L Douglas, PhD, MD, Study Director — THEVAX Genetics Vaccine
Locations (11):
- United States (11):
  - Visions Clinical Research - Tucson, Tucson, Arizona
  - Red Rocks OBGYN, Lakewood, Colorado
  - Progressive Medical Research, Port Orange, Florida
  - Comprehensive Clinical Trials, LLC, West Palm Beach, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - ProHEALTH Care Associates LLP, Port Jefferson, New York
  - Unified Women's Clinical Research, Raleigh, North Carolina
  - Unified Women's Clinical Research, Winston-Salem, North Carolina
  - Complete Healthcare for Women, Columbus, Ohio
  - Penn Fertility Care/Reproductive Research Unit Univ of Pennsylvania, Philadelphia, Pennsylvania
  - Insearch-Tidewater Clinical Research, Norfolk, Virginia